CLINICAL TRIAL: NCT05017363
Title: Evaluation of Effectiveness of Child-oriented Goal-setting in Paediatric Rehabilitation (the ENGAGE Approach): A Pragmatic Cluster Randomized Controlled Trial and Economic Analysis
Brief Title: Evaluation of the Effectiveness of Child-oriented Goal-setting in Paediatric Rehabilitation (the ENGAGE Approach)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RES0044126
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Neurodevelopmental Disorders
Keywords: Goal-setting; Children; Engagement in Therapy
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — engage 8200

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (ENGAGE) (Experimental): Therapists will consist of pairs within sites providing similar interventions to similar children so that treatment and child characteristics other than the goal-setting intervention will be similar within each site. Therapists will use principles-based goal-setting approaches and strategies in the goal-setting toolbox. It is anticipated that treatment block lengths will vary from 3-8 sessions over 2-8 weeks, representing typical clinical variation.
  Interventions: Procedure: ENGAGE
- Usual Care Group (Control) (No Intervention): The control group will comprise usual care.

INTERVENTIONS:
Procedure: ENGAGE — Goal-setting approach and strategies including the Perceived Efficacy and Goal Setting Tool (PEGS), which is established goal setting tools for children aged 5-9. Administration of the Canadian Occupational Performance Measure (COPM), the most widely used goal-setting tool in paediatric rehabilitation that has been used with children as young as seven years. Introducing simple strategies to assist children in identifying goals and to ensure ongoing focus on goals using principles of motivational interviewing, strategies to assess and nurture perceived competence (self-efficacy), and child-friendly feedback strategies on goal-related performance.
  Arms: Intervention Group (ENGAGE)

SUMMARY:
Children with disabilities often access rehabilitation services to improve their abilities to participate in everyday activities. Goal-directed therapy is considered an important therapeutic strategy to achieve outcomes that are meaningful to families. Not a lot is known about the effects of goal setting on rehabilitation outcomes. Strategies to help children participate in the goal-setting process are rarely used in clinical practice. The aim of this project is to test the effects of a child-focussed goal-setting approach, Enhancing Child Engagement in Goal Setting (ENGAGE), on therapy outcomes. The investigators are also interested in service use and the cost vs. benefits of the ENGAGE approach compared to usual practice. Children with neurodevelopmental disabilities aged 5-12 years old (n=96) who access paediatric rehabilitation services at six rehabilitation sites will participate. Therapists (n=24) at participating sites will be randomized into 1) the ENGAGE intervention group or 2) the usual therapy practice control group. Children will participate in the ENGAGE approach to goal setting or usual practice based on the allocation of their therapist. The investigators will determine if the ENGAGE approach to goal setting affects child goal performance, satisfaction with goal performance, functional abilities, participation, and parent and child quality of life. The investigators will also evaluate differences in parent and child quality of life in relation to parent costs (e.g., absenteeism, presenteeism, travel costs) and compare amount of therapy time between the two groups to see which approach is more cost-effective and efficient. The investigators will also ask children, parents, therapists, and managers to discuss aspects that influenced effective implementation of the ENGAGE approach. This study could provide evidence to improve meaningful child and family outcomes in paediatric rehabilitation and improve the efficiency of paediatric rehabilitation services.

DETAILED DESCRIPTION:
PURPOSE:

This pragmatic trial aims to improve health outcomes for children with neurodevelopmental disabilities (NDD) using a novel therapist-targeted, theory-driven, evidence-based approach to goal setting, the Enhancing Child Engagement in Goal Setting (ENGAGE) approach. This study includes an economic analysis and service utilization component and an implementation process analysis to evaluate cost-effectiveness and to support long-term sustainability.

RESEARCH QUESTIONS:

Primary question: Does ENGAGE improve children's engagement in therapy, goal-related performance (primary outcome), functional abilities, participation in home, school and/or community, and child and caregiver quality of life compared to the current standard of care?

Secondary questions: 1) What goal, child, family and therapist factors mediate and/or moderate the effects of ENGAGE on the above intervention outcomes? and 2) Does ENGAGE improve cost effectiveness from the perspectives of parents and service delivery efficiency compared to the current standard of care?

METHODOLOGY/IMPLEMENTATION STRATEGY AND EVALUATION:

Study design: This study will use a pragmatic, cluster randomized controlled trial (RCT) design with therapists randomized to one of two groups; the ENGAGE intervention group or the usual care control group. The RCT will be a six-site trial with two groups (ENGAGE training absent/present) with two periods of post-intervention assessment (immediate post-treatment and 3-month follow-up). The trial will take place within established public paediatric rehabilitation sites in Alberta. An economic analysis consisting of a cost-benefit analysis from the perspectives of parents and a comparison of service utilization costs will be conducted in conjunction with the RCT. To facilitate more widespread implementation, a qualitative process evaluation will be conducted to delineate core versus peripheral components of the intervention, and therapist, child and parent perspectives on the contextual features that influenced implementation.

Sample: The sample size will be 96 children (12 therapists as clusters per group and 4 children per therapist) at six sites. Based on the pilot work, it is anticipated that child dropout from the pre-post intervention period will be minimal (i.e., less than 5%). A target change score of 2.0, a clinically significant change on the COPM (primary outcome), with a standard deviation of 2.75 corresponds to an effect size of 0.723 for the comparison of means. A sample size of 96 will enable us to detect an effect size of at least 0.682 in the primary outcome (COPM performance rating) with alpha=0.05 and 80% power assuming an intra-cluster correlation (ICC) of 0.1 using a two-sided, cluster adjusted, t-test for the comparison of means. The investigators have selected an ICC of 0.1 based on results of a previous cluster RCT with children with cerebral palsy (ICCs between 0.08 to 0.13). Since therapist attrition is possible over the duration of the study, the investigators have designed the sampling strategy so that a cluster size of 11 would still provide 80% power to detect an effect size of 0.716, below our target effect size. Smaller effect sizes will be detectable if the ICC is smaller than 0.1. The sample size has been adjusted from 88 to 96 to allow for an 8% loss to follow-up (1 therapist, 4 children per group). The investigators do not anticipate retention issues for the baseline and post-intervention assessments (primary evaluation period). The probability of loss to follow-up may increase at the 3-month follow-up assessment. Our estimate of loss to follow-up is based on our experience with trials with children with disabilities.

Recruitment: Over 18 months, children (n=96) will be sequentially recruited by 24 therapists from six paediatric Alberta rehabilitation sites (4 children per therapist). The investigators have confirmed partner sites, who believe these numbers are feasible based on the number of therapists and typical caseloads in their programs and our previous experience collecting pilot data. Study therapists will identify potential participants who they are about to see for regular therapy. Therapists will provide families with a tablet with a video of the researchers introducing the study and inviting them to participate (see video script in documentation section), or they will email the video link to families who are receiving services virtually due to COVID 19 restrictions. Parents can either consent to participate through an online form (REDCap) or request additional information by signing the contact information form. Contact information will be provided to the researchers if parents sign either of these two forms. If parents request additional information, they will be contacted and if they are interested in participating after a discussion about the study, consent will obtained (audio-recorded). Child assent will be obtained by the treatment therapist at the next therapy visit or will be obtained over the phone as well. The investigators will use the most feasible option as suggested by parents. Some children will not be able to verbalize assent over the telephone. If parents do not wish to participate, treatment with their therapists, will continue as usual.

Randomization: A computer-generated, permuted-block randomization sequence using site as a stratification variable will be used to allocate 24 OTs and PTs across 6 sites to the ENGAGE or control group to ensure balanced groups. Blocked randomization by site will facilitate consistency of therapy interventions and child characteristics between groups with the exception of the ENGAGE in the intervention arm. If therapists within more than one program at a site participate, therapists will also be randomized by program. The randomization sequence will be uploaded to REDCap to allow for centralized, online randomization. Randomization of therapists (and not children) will decrease contamination in the usual practice group (i.e., so therapists are not asked to go between intervention and usual care practices) and blocking by site will facilitate equal group distribution related to therapy interventions (e.g., types of therapy) and child characteristics (e.g., age, diagnosis). Dr. Rosychuk (co-applicant) will generate the randomization sequence and an independent research assistant not associated with the trial will conduct blinded randomization.

Study groups: Intervention Group - Therapists will receive training on our principles-based goal setting approach and strategies in the goal setting toolbox. Training will include an overview of tools and strategies including the Perceived Efficacy and Goal Setting Tool (PEGS), which is an established goal setting tool for children aged 5-9. In addition, training will be provided on administration of the Canadian Occupational Performance Measure (COPM), the most widely used goal setting tool in paediatric rehabilitation that has been used with children as young as seven years. The investigators will introduce simple strategies to assist children in identifying goals and to ensure ongoing focus on goals using principles of motivational interviewing, strategies to assess and nurture perceived competence (self-efficacy), and child-friendly feedback strategies on goal-related performance. Therapists will consist of pairs within sites providing similar interventions to similar children so that treatment and child characteristics other than the goal setting intervention will be similar within each site.

Control group - The control group will comprise usual care. Research on goal setting in paediatric rehabilitation in Alberta suggests that usual practice is highly variable, often reflecting therapist preference and a lack of formalized goal setting processes. Research conducted elsewhere also suggests that rehabilitation goals are inconsistently established and documented and not based on theoretically informed principles. Recent findings from our pilot work revealed that adherence to our four principles was a significant shift from traditional practice that did not emphasize child engagement, attention to self-efficacy, or strategies based on principles of behaviour change.

Treatment duration and intensity for both groups will differ based on nature of goals, treatment strategies, and family preference. It is anticipated that treatment block lengths will vary from 3-8 sessions over 2-8 weeks, representing typical clinical variation.

Fidelity monitoring- Following the training, the investigators will track the strategies used by ENGAGE therapists to evaluate treatment fidelity prior to recruiting participants. Feedback will be provided as needed to therapists as part of the implementation plan to facilitate ongoing and consistent use of the intervention strategies. This feedback will be provided through email, phone or Zoom. Treatment frequency, intensity, intervention strategies, and feedback frequency and mechanisms will be documented by therapists at each treatment session. Co-interventions will be monitored for each participant. Recruitment and formalized data collection will begin once intervention therapists at the site achieve an acceptable level of fidelity defined as adherence to ENGAGE principles at least 90% of the time. For example, the investigators will monitor the extent children are involved in identifying their own goals and how often therapists use feedback on goal-related performance at each treatment session. Practices will also be monitored in the control group using an open-ended form to prevent contamination from exposure to ENGAGE principles. Ongoing documentation of practices and monitoring will be used to evaluate the need for additional or different implementation support in the intervention group and to enable comparison of group practices.

Data collection: Identical assessments will be conducted at 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment. Three months is a common time period for follow-up for rehabilitation intervention studies reflecting retention within a time frame reasonable to attribute to the intervention. Trained assessors, blinded to group allocation, will complete the measures with families using Zoom to account for risks associated with COVID-19. The investigators will email a copy of all tools to each family, and screen share the same tools using Zoom to go through with the family and document answers. Family members will be blinded to all initial responses on the measures. It is hypothesized significant between group differences in favour of the intervention group on the primary and secondary outcomes. The investigators hypothesize that these differences will be maintained at follow-up across measures. All outcome measures will be used at baseline, post-intervention and at 3-month follow-up, administered by trained assessors blinded to group allocation. All outcome measures are established tools, and have strong psychometric properties with children with disabilities and/or their parents.

An economic analysis consisting of a cost benefit analysis from the family perspective will be conducted in conjunction with this trial. Costs related to ENGAGE relative to typical care will be tracked using a therapy session questionnaire for both groups. In addition, total costs incurred per child during the intervention will be determined by multiplying therapist direct and indirect (e.g., documentation) time by a corresponding unit price. Mean cost per child will then be calculated for each group. Costs from the family perspective will be tracked using a parent questionnaire and outcomes will be parent and child quality of life (CarerQol-7D and KIDSCREEN-10).

Analysis: Data and demographic characteristics will be described (e.g., means, standard deviations) for both groups. Change scores (post minus pre, follow-up minus post) will be summarized for each outcome, with COPM-P changes post intervention as the primary analysis (Question 1) and the other outcomes as secondary analyses. For each change score and outcome, a cluster adjusted t-test will be used to compare mean change score between groups (ENGAGE, control). A confidence interval will be reported for the difference between group mean scores. Mixed effects linear regression models on all outcomes will include group and time (fixed effects), a therapist random effect (to adjust for the clustering), and a child random effect (to adjust for repeated measures on each child). Time will be a categorical variable so that post and follow-up times can be compared with pre-treatment assessments. A time by group interaction will also be considered to assess the effects of group.

Question 2: Mixed effects multiple linear regression models similar to the above will also be developed for each outcome with the additional variables of site, site by group as an interaction (to assess site effect) and other theoretically important variables (e.g., cognitive abilities, age, parenting style) as covariates. Variables will be dropped from the model one at a time if the p-value is <0.05 and not needed for model fit. This modelling will allow us to assess the effects of the interventions in the presence of important variables that may not be balanced across groups by randomization. This approach will be used since there may be some systematic differences in therapist caseload. All main analyses will be based on 'as per protocol' analysis, as recommended for pragmatic trials. Analyses will be performed by an analyst blinded to group assignment using R, directed by Dr. Rosychuk.

Question 3: Mean cost per child and the mean effectiveness result per child for each group will be represented in an incremental cost-effectiveness ratio (ICER) - the ratio of the difference between groups in mean cost per patient to the difference in mean effectiveness using the two quality of life measures (CarerQol and KIDSCREEN) as outcomes. Extensive sensitivity analysis including probabilistic sensitivity analysis will be undertaken to test robustness of the results.

Process evaluation: Data collection will occur pre-implementation, during and post-implementation, as outlined below.

Pre-implementation: Quantitative data: Therapists will complete the readiness for change scale of the Organizational change questionnaire - Climate of Change, Processes, and Readiness measure at the training session for ENGAGE. Therapists and managers will complete a short demographic questionnaire.

Qualitative data: As part of their training, therapists in the ENGAGE group will discuss anticipated barriers to this approach as well as potential strategies to optimize implementation. This discussion will be very informal and facilitated by broad discussion questions. Front-line managers will also participate in 45-minute interviews (either over the phone or Zoom depending on what is most convenient). These interviews will be designed to understand the managers' anticipated barriers to the ENGAGE approach. All interviews will be audio-recorded and professionally transcribed.

During implementation: Bi-weekly meetings will be conducted over Zoom with the therapists at each site. These interviews will be conducted by phone or Zoom, based on participant preference. The purpose of these discussions will be to regularly assess and document barriers and facilitators to implementation. The discussion will be very informal and informed by the Consolidated Framework for Implementation Research (CFIR) and the Theoretical Domains Framework (TDF). These discussion will be audio-recorded and transcribed.

Post-implementation: Qualitative data: Semi-structured interviews will be conducted post-implementation with both the parent and child-participants (ENGAGE condition), therapists (ENGAGE condition) and managers. Parent and child-participants will be interviewed before or following their post-implementation assessment. Therapists allocated to the ENGAGE group will be interviewed individually either over the phone/video following the completion of therapy (within 14 days). Managers will be interviewed shortly after all of their therapists have completed the study. CFIR framework was used in conjunction with the TDF to develop the interview guides. Interviews (45-60 minutes) will be audio-recorded and professionally transcribed.

Data will be analyzed using inductive thematic analysis following Braun & Clarke's 6-phase framework. Demographic data and the questionnaire data (readiness for change) from the therapist will be will be summarized using descriptive statistics. Journaling will be used to record preliminary themes/ideas about the data, experiences in the research process and rationale for data collection and analysis decisions, and to facilitate researcher reflexivity.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Physical Therapy and/or Occupational Therapy for a period of direct treatment,
* English speaking

Exclusion Criteria:

* Presence of a progressive condition
* The child has uncontrolled seizures (i.e., had a seizure within the past 2 months).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Self-perceived, goal-related performance on the COPM (COPM-P) | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment.
  Canadian Occupational Performance Measure, Performance rating, 1 (not able to do it -10 able to do it extremely well).

SECONDARY OUTCOMES:
Participation | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment
  Participation and Environment Measure for Children & Youth (PEM-CY)
Child Quality of Life | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment
  Child Quality of Life KIDSCREEN-10
Parent Quality of Life | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment
  Parent Quality of Life: Caregiver Quality of Life (CarerQol-7D)
Functional Abilities | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment
  Pediatric Evaluation of Disability Inventory (PEDI-CAT)

OTHER OUTCOMES:
Child engagement in therapy | At each treatment session (session frequency will vary; estimated # of sessions is 3-10. )
  Pediatric Rehabilitation Intervention Measure of Engagement (Service Provider version)(PRIME-SP)
Mastery Motivation | Baseline
  Dimensions of Mastery Children's Motivation Questionnaire-18
Parenting style | Baseline
  Parenting Behaviours and Dimensions Questionnaire
Autonomy | Change from baseline (pre-treatment) to post-treatment (within 10 days), and change between post-treatment and 3-months post-treatment
  Likert Scale (1-10; 10 indicates high level of autonomy)
Perceived Competence | baseline
  Belief in Goal Self-Competence Scale (BiGSS) (1-10; 10 indicates high level of perceived competence)
Child-rated experience measure of practitioner empathy | post-treatment (within 10 days)
  Visual CARE

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Pritchard, PhD, Principal Investigator — University of Alberta; Sandra Hodgetts, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Pritchard-Wiart L, Thompson-Hodgetts S, McKillop AB, Rosychuk R, Mrklas K, Zwaigenbaum L, Zwicker J, Andersen J, King G, Firouzeh P. A multi-center, pragmatic, effectiveness-implementation (hybrid I) cluster randomized controlled trial to evaluate a child-oriented goal-setting approach in paediatric rehabilitation (the ENGAGE approach): a study protocol. BMC Pediatr. 2022 Jun 29;22(1):375. doi: 10.1186/s12887-022-03381-4. PMID 35764983